CLINICAL TRIAL: NCT02705443
Title: Early Identification of Suspected Deep Tissue Injury (sDTI) Utilizing Long-Wave Thermographic Imaging (LWIT)
Brief Title: Early Identification of Suspected Deep Tissue Injury (sDTI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wound Vision (Industry)
Responsible Party: Sponsor
Other Study IDs: WV15CL-0001
Record Dates: First submitted 2016-03-02; First posted 2016-03-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Pressure Ulcer; Bed Sore
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Tissue w/ Thermographic Anomaly: * Visibly undamaged tissue with anomaly identified by the thermographic image
  * No intervention
  * Standard of care
  Interventions: Other: No Intervention
- Tissue w/o Thermographic Anomaly: * Visibly undamaged tissue with no anomaly identified by the thermographic image
  * No intervention
  * Standard of care
  Interventions: Other: No Intervention
- Tissue w/ Visible Anomaly: * Visibly damaged tissue
  * No intervention
  * Standard of care
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Standard of Care Only

SUMMARY:
The purpose of this study is to further clarify existing research on the early identification and documentation of suspected deep tissue injury (sDTI). Basic principles of physiology along with prior research suggests that sDTI has quantifiable amounts of heat (or lack thereof) relative to surrounding tissue that will exhibit characteristic thermal signatures (temperature). These signatures will be measured and quantitatively recorded using long-wave infrared thermography (LWIT) to not only identify sDTI, but to also learn more about their pathophysiological evolution. Additionally, the LWIT physiological data will be cross-compared to the gold standard of visual assessment and other current standards of wound evaluation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Can tolerate position changes ≥ 10 minutes
* Non-pregnant

Exclusion Criteria:

* Therapies/treatments cannot be safely suspended to for an imaging session
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects admitted to a long-term acute care hospital (LTACH).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of anatomical areas with intact skin and a thermographic anomaly that progress to a stageable pressure ulcer | Up to 25 days
  Sensitivity and specificity of a thermographic anomaly that progresses to a stageable pressure ulcer
Number of anatomical areas with intact skin and a thermographic anomaly that do not progress to a stageable pressure ulcer | Up to 25 days
  Sensitivity and specificity of a thermographic anomaly that does not progress to a stageable pressure ulcer

SECONDARY OUTCOMES:
Temperature change associated with anatomical areas after a stageable pressure ulcer occurs | Up to 25 days

CONTACTS AND LOCATIONS:
Locations (1):
- Kindred Hospital Dayton, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided